CLINICAL TRIAL: NCT02952222
Title: The Synergistic Effect of Dexmedetomidine on Propofol for Sedation for Pediatric Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keira Mason (Other)
Responsible Party: Sponsor-Investigator, Keira Mason, MD, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00020516
Record Dates: First submitted 2016-03-14; First posted 2016-11-02 (Estimated); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Propofol (Group P) (Active Comparator): Propofol only
  Interventions: Drug: Propofol (Group P)
- Propofol with Dexmedetomidine (Group DP) (Active Comparator): Propofol with Dexmedetomidine
  Interventions: Drug: Dexmedetomidine; Drug: Propofol (Group DP)

INTERVENTIONS:
Drug: Dexmedetomidine — Patients in Group DP will receive 0.5 mcg/kg Dexmedetomidine (DEX) administered over 1 minute followed by an infusion of 0.15 mcg/kg/hr. Following the 0.5 mcg/kg DEX bolus, propofol will be administered with the identical protocol (with same endpoint of Bispectral Index (BIS) 40-50) of the P Group. Propofol infusion will be started at 200 mcg/kg/min and will be titrated throughout the procedure to maintain a BIS 40-50. Propofol may be administered prn in 10-20 mg increments for any abrupt patient movement which may compromise the continuity of the procedure.
  Other Names: Precedex
  Arms: Propofol with Dexmedetomidine (Group DP)
Drug: Propofol (Group P) — Patients in Group P will receive intravenous propofol in bolus increments (2.0 mg/kg bolus over one minute then 0.5 mg/kg bolus q 1 minute titrated to a BIS of 40-50). These patients will be maintained with a continuous intravenous infusion of propofol starting at 200 mcg/kg/min and will be titrated to an endpoint of maintaining a BIS level of 40-50.
  Arms: Propofol (Group P)
Drug: Propofol (Group DP) — Patients in Group DP will receive 0.5 mcg/kg DEX administered over 1 minute followed by an infusion of 0.15 mcg/kg/hr. Following the 0.5 mcg/kg DEX bolus, propofol will be administered with the identical protocol (with same endpoint of BIS 40-50) of the P Group. Propofol infusion will be started at 200 mcg/kg/min and will be titrated throughout the procedure to maintain a BIS 40-50. Propofol may be administered prn in 10-20 mg increments for any abrupt patient movement which may compromise the continuity of the procedure.
  Arms: Propofol with Dexmedetomidine (Group DP)

SUMMARY:
The primary aim of this study is to compare the propofol requirements of children who receive propofol with that of children who receive dexmedetomidine prior to propofol, for sedation for upper and lower endoscopic procedures.

DETAILED DESCRIPTION:
Both propofol and dexmedetomidine may be used to achieve adequate sedation conditions. Propofol has been described to produce successful conditions for completion of the intended study in almost 99% of the patients. However, in a study that reviewed outcomes when using propofol for almost 50,000 pediatric procedures, propofol was associated with stridor, laryngospasm, airway obstruction, wheezing or central apnea at a rate of 1 in 65 sedations. The need for airway and ventilation interventions which include oral/nasal airway placement, positive pressure mask ventilation and tracheal intubation occurred at a rate of 1 in 70 sedations. Hemodynamic and respiratory fluctuations of a minimum of 30% fluctuations in heart rate, blood pressure or respiratory rate occurred at a rate of 1 in 165 sedations. Another recent study cited similar incidences of hemodynamic variability with propofol as well as inhalational anesthesia in the outpatient pediatric setting.

Until 2015, dexmedetomidine had been one of the standard drugs administered for sedation in children who require radiologic diagnostic imaging studies (MRI, CT and Nuclear Medicine) in the Department of Radiology at Boston Children's Hospital (BCH). Over 17,000 infants, children and developmentally compromised young adults had been sedated with dexmedetomidine in BCH without a cardiac or respiratory arrest, or a need to provide positive pressure assisted ventilation.

This study will determine if administration of dexmedetomidine with propofol administration will result in lower doses of the latter, which may mean safer outcomes in sedation for upper and lower endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7-18 years who are scheduled for upper or lower endoscopic procedures at Boston Children's Hospital and meets criteria to receive dexmedetomidine or propofol sedation for upper and lower endoscopic procedures
* Provides written consent to participate in the research study
* For females of childbearing age, pregnancy test is negative

Exclusion Criteria:

* Do not meet established sedation criteria
* Refuses administration of study medication prior to sedation
* History of allergy, intolerance, or reaction to dexmedetomidine or propofol or hypersensitivity
* Current, repaired or risk of Moya-Moya disease
* Recent stroke (cerebrovascular accident) within past 6 months
* Uncontrolled hypertension
* Concomitant use of opioids, beta antagonist, alpha 2 agonist or calcium channel blocker
* Egg, soy or lecithin allergy
* BMI greater than 30 or weight above 110th percentile
* Refuses insertion of intravenous catheter while awake
* Currently receiving pharmacologic agents for hypertension or cardiac disease
* Currently receiving or has received digoxin within the past 3 months
* Active, uncontrolled gastroesophageal reflux - an aspiration risk
* Current (or within past 3 months) history of apnea requiring an apnea monitor
* Unstable cardiac status (life threatening arrhythmias, abnormal cardiac anatomy, significant cardiac dysfunction)
* Craniofacial anomaly, which could make it difficult to effectively establish a mask airway for positive pressure ventilation if needed
* Active, current respiratory issues that are different from the baseline status (pneumonia, exacerbation of asthma, bronchiolitis, respiratory syncytial virus)

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keira Mason, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mason KP, Park RS, Sullivan CA, Lukovits K, Halpin EM, Imbrescia ST, Cavanaugh D, Prescilla R, Fox VL. The synergistic effect of dexmedetomidine on propofol for paediatric deep sedation: A randomised trial. Eur J Anaesthesiol. 2021 May 1;38(5):541-547. doi: 10.1097/EJA.0000000000001350. PMID 33009191

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol (Group P): Propofol only
  Propofol (Group P): Patients in Group P will receive intravenous propofol in bolus increments (2.0 mg/kg bolus over one minute then 0.5 mg/kg bolus q 1 minute titrated to a Bispectral Index (BIS) of 40-50). These patients will be maintained with a continuous intravenous infusion of propofol starting at 200 mcg/kg/min and will be titrated to an endpoint of maintaining a BIS level of 40-50.
- Propofol With Dexmedetomidine (Group DP): Propofol with Dexmedetomidine
  Dexmedetomidine: Patients in Group DP will receive 0.5 mcg/kg DEX administered over 1 minute followed by an infusion of 0.15 mcg/kg/hr. Following the 0.5 mcg/kg Dexmedetomidine (DEX) bolus, propofol will be administered with the identical protocol (with same endpoint of BIS 40-50) of the P Group. Propofol infusion will be started at 200 mcg/kg/min and will be titrated throughout the procedure to maintain a BIS 40-50. Propofol may be administered prn in 10-20 mg increments for any abrupt patient movement which may compromise the continuity of the procedure.
  Propofol (Group DP): Patients in Group DP will receive 0.5 mcg/kg DEX administered over 1 minute followed by an infusion of 0.15 mcg/kg/hr. Following the 0.5 mcg/kg DEX bolus, propofol will be administered with the identical protocol (with same endpoint of BIS 40-50) of the P Group. Propofol infusion will be started at 200 mcg/kg/min and will be titrated throughout the procedure to maintain a BIS 40-50. Propofol may be administered prn in 10-20 mg increments for any abrupt patient movement which may compromise the continuity of the procedure.
Period: Overall Study
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
Started | 19 | 20
Completed | 16 | 19
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Propofol With Dexmedetomidine (Group DP): Propofol with Dexmedetomidine
  Dexmedetomidine: Patients in Group DP will receive 0.5 mcg/kg DEX administered over 1 minute followed by an infusion of 0.15 mcg/kg/hr. Following the 0.5 mcg/kg DEX bolus, propofol will be administered with the identical protocol (with same endpoint of BIS 40-50) of the P Group. Propofol infusion will be started at 200 mcg/kg/min and will be titrated throughout the procedure to maintain a BIS 40-50. Propofol may be administered prn in 10-20 mg increments for any abrupt patient movement which may compromise the continuity of the procedure.
  Propofol (Group DP): Patients in Group DP will receive 0.5 mcg/kg DEX administered over 1 minute followed by an infusion of 0.15 mcg/kg/hr. Following the 0.5 mcg/kg DEX bolus, propofol will be administered with the identical protocol (with same endpoint of BIS 40-50) of the P Group. Propofol infusion will be started at 200 mcg/kg/min and will be titrated throughout the procedure to maintain a BIS 40-50. Propofol may be administered prn in 10-20 mg increments for any abrupt patient movement which may compromise the continuity of the procedure.
- Total: Total of all reporting groups
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP) | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 20 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (2.9) | 14.4 (3.2) | 13.9 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 13 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 19 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Propofol Requirements With Pre-treatment of Dexmedetomidine With Children Who do Not Receive Dexmedetomidine.
Description: Compare the total propofol requirements (in mg/kg/min) of children who receive intravenous propofol with pre-treatment of dexmedetomidine with the propofol requirements in children who do not receive dexmedetomidine.
Time Frame: up to 3 hours
Measure: Median (Inter-Quartile Range); unit: mg/kg/min
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
Number analyzed (Participants) | 16 | 19
mg/kg/min | 0.4 [0.2 to 0.5] | 0.23 [0.1 to 0.5]

2. Secondary Outcome: Frequency of Adverse Events and the Need for Airway Interventions
Description: To compare propofol to dexmedetomidine with respect to the frequency of adverse events and the need for airway interventions
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
Number analyzed (Participants) | 16 | 19
Participants | 0 | 1

3. Secondary Outcome: Time Required to Achieve Sedation
Description: To compare propofol to dexmedetomidine with respect to the time required to receive sedation
Time Frame: up to 30 minutes
Measure: Mean (Full Range); unit: minutes
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
Number analyzed (Participants) | 16 | 19
minutes | 7.5 [3 to 14] | 7 [3 to 12]

4. Secondary Outcome: Time Required to Meet Discharge Criteria From Recovery Room
Description: To compare the propofol-only group to dexmedetomidine-propofol group with respect to the time required to meet discharge criteria from recovery room
Time Frame: up to 4 hours
Measure: Mean (Full Range); unit: minutes
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
Number analyzed (Participants) | 16 | 19
minutes | 63 [46 to 91] | 60 [20 to 121]

5. Secondary Outcome: Adverse Events
Description: To compare the propofol-only group to dexmedetomidine-propofol group with respect to adverse events
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
Number analyzed (Participants) | 16 | 19
Participants | 0 | 1

6. Secondary Outcome: Number of Unplanned Airway Interventions According to the World Society of Intravenous Anaesthesia (SIVA) Adverse Sedation Event Reporting Tool
Description: To compare the propofol-only group to dexmedetomidine-propofol group with respect to the need for unplanned airway interventions
Time Frame: up to 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
Number analyzed (Participants) | 16 | 19
Participants | 0 | 1

7. Secondary Outcome: Emergence Delirium
Description: To compare the propofol-only group to dexmedetomidine-propofol group with respect to the Pediatric Anesthesia Emergence Delirium (PAED) score. The PAED is a scale that measures emergence delirium in children and adolescence as they wake up from anesthesia. The lowest achievable score is 0 and is consistent with no emergence delirium (best outcome). The highest achievable score is 20 and is consistent with emergence delirium (worse outcome).
Time Frame: up to 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
Number analyzed (Participants) | 16 | 19
Participants
  Score>=10 | 15 | 18
  Score<10 | 1 | 1

8. Secondary Outcome: Time to BIS Score
Description: To compare the propofol-only group to dexmedetomidine-propofol group with respect to time (in minutes) of return of BIS score to baseline (pre-sedation level) in recovery room
Time Frame: up to 6 hours
Measure: Mean (Full Range); unit: minutes
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
Number analyzed (Participants) | 16 | 19
minutes | 45 [35 to 53] | 50 [26 to 54]

9. Secondary Outcome: Duration of Sedation
Description: To compare the propofol-only group to dexmedetomidine-propofol group with respect to the duration of sedation
Time Frame: up to 3 hours
Measure: Mean (Full Range); unit: minutes
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
Number analyzed (Participants) | 16 | 19
minutes | 22 [10 to 72] | 33 [10 to 93]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each patient for up to 3 days, starting from the time of first drug administration (DEX or propofol).
Arm/Group | Propofol (Group P) | Propofol With Dexmedetomidine (Group DP)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 0/16 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol (Group P) (N=16) | Propofol With Dexmedetomidine (Group DP) (N=19)
Question of Bronchospasm and laryngospam (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Oxygen desaturation (75 to 90%) for less than 60s, requiring two interventions: additional sedative was administered (minimal risk) and bag-valve mask-assisted ventilation (moderate risk). No other unintended events occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT02952222/Prot_SAP_000.pdf